CLINICAL TRIAL: NCT05232383
Title: Benefits and Risks of Artificial Light Exposure: Characterisation of Effects on Alertness, Sleep, Cognitive Performance, Mood and Biological Rhythms
Acronym: LumEnColor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8076
Record Dates: First submitted 2021-01-18; First posted 2022-02-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Human Sleep and Chronobiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Wp (Active Comparator)
  Interventions: Device: polychromatic light
- Wn (Active Comparator)
  Interventions: Device: polychromatic light
- Gn (Active Comparator)
  Interventions: Device: green light
- Gp (Active Comparator)
  Interventions: Device: green light
- Rp (Active Comparator)
  Interventions: Device: red light
- Rn (Active Comparator)
  Interventions: Device: red light

INTERVENTIONS:
Device: polychromatic light — Application of polychromatic light at different times of day
  Arms: Wp
Device: polychromatic light — Application of polychromatic light for 2h30 at different times of day with sleep
  Arms: Wn
Device: red light — Application of red light at different times of day
  Arms: Rp
Device: red light — Application of red light at different times of day with sleep
  Arms: Rn
Device: green light — Application of green light at different times of day
  Arms: Gp
Device: green light — Application of green light at different times of day with sleep
  Arms: Gn

SUMMARY:
The purpose of this project is to study the influence of light on sleep, wakefulness, EEG activity and cognitive performances.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18 to 40 years
* With a hint of Bodymass index (BMI) between 17 and 30 kg.m - 2
* healthy subject determined by a clinical examination, a psychological interview, a blood test, a urine analysis
* Subject with a score<6 questionnaire PSQI ("Sleep Questionnaire Pittsburgh")
* Subject agreeing to maintain a regular sleep/wake rhythm during the study
* Subject agreeing to refrain from caffeine, nicotine, alcohol, psychotropic drugs, cannabis or other drugs, during the study
* Signed informed consent
* Subjectaffiliated to a social protection scheme

Exclusion Criteria:

* somatic diseases: cardiovascular, respiratory, gastrointestinal, hematopoietic, Visual
* immune system diseases
* kidneys and urinary tract diseases
* endocrine and metabolic diseases
* neurological diseases
* infectious diseases
* thrombocytopenia or other malfunction of blood platelets
* Subject with risk of thrombosis, including subject with a history of phlebitis, smoker under oral contraceptive...
* Subject with an addiction to caffeine, nicotine, alcohol, psychotropic drugs, cannabis, or any other drug
* Subject treatment contraindicated or inadvisable in combination with heparin
* blood donation in the previous 3 months before the inclusion
* Participation in other clinical trials
* Work by shifts in the year preceding the inclusion
* Trans-meridian travel (> 2 time zones) in the month previous the inclusion
* Impossibility to give enlightened information (subject in an emergency situation, understanding difficulties,...)
* Subject under safeguard of justice
* Subject under tutorship or curatorship
* Pregnancy (women of childbearing age)
* Breastfeeding
* Diet incompatible with the study's snack choices

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive performances assessed using N-back tasks | up to 56 hours
  N-Back-Task 1, 2, 3
Cognitive performances assessed using Psychomotor Vigilance task (PVT) | up to 56 hours
  Psychomotor Vigilance task (PVT)
Cognitive performances assessed using Paced Visual Serial Addition Task (PVSAT) | up to 56 hours
  Paced Visual Serial Addition Task (PVSAT)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice BOURGIN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No